CLINICAL TRIAL: NCT03737734
Title: A Safety and Effectiveness Study of Intratumoral Diffusing Alpha Radiation Emitters for the Treatment of Malignant Cutaneous, Mucosal or Superficial Soft Tissue Neoplasia
Brief Title: Alpha Radiation Emitters Device for the Treatment of Cutaneous, Mucosal or Superficial Soft Tissue Neoplasia (DaRT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-CMN-02
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-11

CONDITIONS: Skin Cancer; Mucosal Neoplasm of Oral Cavity; Soft Tissue Neoplasm
Keywords: Squamous Cell Carcinoma; SCC; Skin Cancer; Skin metastasis; HNSCC; Carcinoma, Squamous; CMN; Basal cell carcinoma; Superficial sarcoma; Kaposi sarcoma; Alpha radiation; Cutaneous lesion; Tongue cancer; Lip cancer; Brachytherapy
MeSH Terms: conditions — Skin Neoplasms; Soft Tissue Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Basal Cell; Sarcoma, Kaposi; Tongue Neoplasms; Lip Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of a seed(s), loaded with Radium-224, securely fixed in the seeds. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.
  Other Names: DaRT

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for superficial cutaneous, mucosal or soft tissue neoplasia

DETAILED DESCRIPTION:
This will be a prospective, open label, single arm, controlled study, assessing the safety and efficacy of diffusing alpha emitters radiation therapy (DaRT) delivered through radioactive seeds inserted into the tumor.

This approach combines the advantages of local intratumoral irradiation of the tumor, as used in conventional brachytherapy, with the power of the alpha radiation emitting atoms, that will be introduced in quantities considerably lower than radiation therapy already used in patients.

Superficial lesions with histopathological confirmation of malignancy will be treated using DaRT seeds.

Reduction in tumor size 70 days after DaRT insertion will be assessed. Safety will be assessed by the incidence, severity and frequency of all Adverse Events (AE).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histopathological confirmation of primary or secondary malignant cutaneous neoplastic lesions, or oral cavity mucosal tumors, or superficial soft tissue sarcoma.
* Subjects with a tumor size ≤ 7 centimeters in the longest diameter.
* Patients who have either failed first-line treatment, or are medically unfit for standard of care (surgery, external-beam radiation therapy or chemotherapy), or refuse standard of care.
* Subjects' ECOG Performance Status Scale is < 2.
* Subjects' life expectancy is more than 6 months.
* Platelet count ≥100,000/mm3.
* International normalized ratio of prothrombin time ≤1.8.
* Creatinine ≤1.9 mg/dL.
* Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test.
* Subjects are willing to sign an informed consent form.

Exclusion Criteria:

* Subject has a tumor of Keratoacanthoma histology.
* Patients with significant comorbidities that the treating physician deems may conflict with the endpoints of the study (e.g., poorly controlled autoimmune diseases, vasculitis, etc.)
* Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
* High probability of protocol non-compliance (in opinion of investigator)
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Tumor response to DaRT | 9-11 weeks post DaRT insertion
  Assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1)
Adverse Events | Up to 24 Months
  The incidence, frequency, severity and causality of acute adverse events related to the DaRT treatment according to Common Terminology and Criteria for adverse events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Reduction in tumor volume | 9-11 weeks post DaRT insertion
  based on imaging
DaRT seeds placement | Day of insertion procedure
  Assessment by localization of the DaRT seeds in the tumor using CT imaging on the day of DaRT insertion
Change in quality of life | Day 15, Day 30, Day 70, Day 180 post DaRT insertion
  Assessment of patient reported health-related Quality of Life outcome after DaRT, using QoL questionnaire Skindex-16 questionnaire score
Change in quality of life | Day 30, Day 70, Day 180 post DaRT insertion
  Assessment of patient reported health-related Quality of Life outcome after DaRT, using QoL questionnaire Skin Cancer Index (SCI) questionnaire score
Adverse Events | Up to 24 Months
  All Adverse Events (AE) related and unrelated to the study treatment
Progression Free Survival | 24 months post DaRT insertion
  Time elapsed from response to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Noga Kurman, MD, Principal Investigator — Davidof Cancer Institution at Rabin Medical Center Israel
Locations (1):
- Davidof Cancer Institution at the Rabin Medical Center Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No